CLINICAL TRIAL: NCT03184064
Title: Acute Effects of Blackcurrant and Citrus Polyphenol Extracts on Postprandial Glycaemia: The Glu-FX Study
Brief Title: Acute Effects of Blackcurrant and Citrus Polyphenol Extracts on Postprandial Glycaemia
Acronym: Glu-FX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucozade Ribena Suntory (Industry)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HVS-007
Record Dates: First submitted 2017-05-23; First posted 2017-06-12 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Postprandial Period
Keywords: Blackcurrant; Citrus; Polyphenols; Glucose; Postprandial; Metabolism

STUDY DESIGN:
Intervention Model Description: Incomplete block cross-over design. Each participant receives placebo plus 3 out of 4 active treatments.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment arm 1 (Experimental): Participants will receive the placebo, blackcurrant extract (low dose), blackcurrant extract (high dose), citrus extract (low dose) at 4 separate study visits, in a random order. Visits will be separated by at least 7 days.
  Interventions: Dietary Supplement: Blackcurrant extract (low dose); Dietary Supplement: Placebo; Dietary Supplement: Citrus extract (low dose); Dietary Supplement: Blackcurrant extract (high dose)
- Treatment arm 2 (Experimental): Participants will receive the placebo, citrus extract (low dose), blackcurrant extract (high dose), blackcurrant and citrus extracts (low dose / low dose) at 4 separate study visits, in a random order. Visits will be separated by at least 7 days.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Citrus extract (low dose); Dietary Supplement: Blackcurrant extract (high dose); Dietary Supplement: Blackcurrant and citrus extracts (low dose / low dose)
- Treatment arm 3 (Experimental): Participants will receive the placebo, blackcurrant extract (low dose), blackcurrant extract (high dose), blackcurrant and citrus extracts (low dose / low dose) at 4 separate study visits, in a random order. Visits will be separated by at least 7 days.
  Interventions: Dietary Supplement: Blackcurrant extract (low dose); Dietary Supplement: Placebo; Dietary Supplement: Blackcurrant extract (high dose); Dietary Supplement: Blackcurrant and citrus extracts (low dose / low dose)
- Treatment arm 4 (Experimental): Participants will receive the placebo, blackcurrant extract (low dose), citrus extract (low dose), blackcurrant and citrus extracts (low dose / low dose) at 4 separate study visits, in a random order. Visits will be separated by at least 7 days.
  Interventions: Dietary Supplement: Blackcurrant extract (low dose); Dietary Supplement: Placebo; Dietary Supplement: Citrus extract (low dose); Dietary Supplement: Blackcurrant and citrus extracts (low dose / low dose)

INTERVENTIONS:
Dietary Supplement: Blackcurrant extract (low dose) — Participants will consume a small beverage that contains blackcurrant extract (low dose) immediately before a high-carbohydrate meal.
  Arms: Treatment arm 1; Treatment arm 3; Treatment arm 4
Dietary Supplement: Placebo — Participants will consume a small beverage that contains no fruit extracts immediately before a high-carbohydrate meal.
Dietary Supplement: Citrus extract (low dose) — Participants will consume a small beverage that contains citrus extract (low dose) immediately before a high-carbohydrate meal.
  Arms: Treatment arm 1; Treatment arm 2; Treatment arm 4
Dietary Supplement: Blackcurrant extract (high dose) — Participants will consume a small beverage that contains blackcurrant extract (high dose) immediately before a high-carbohydrate meal.
  Arms: Treatment arm 1; Treatment arm 2; Treatment arm 3
Dietary Supplement: Blackcurrant and citrus extracts (low dose / low dose) — Participants will consume a small beverage that contains blackcurrant and citrus extracts (low dose / low dose)immediately before a high-carbohydrate meal.
  Arms: Treatment arm 2; Treatment arm 3; Treatment arm 4

SUMMARY:
Large postprandial glucose responses are associated with increased risk of chronic diseases, including diabetes and cardiovascular disease. Our group have previously shown that fruit polyphenol extracts, when consumed immediately before a mixed carbohydrate meal, reduce postprandial glycaemia. The aim of this study is to investigate the effects of a blackcurrant polyphenol extract and citrus polyphenol extract (and their combination), on postprandial glycaemia, insulinaemia and gastrointestinal hormone concentrations following a mixed carbohydrate test meal. It is hypothesised that blackcurrant and citrus extracts alone will inhibit glycaemia compared to placebo, and a combination of the two will have a greater effect.

DETAILED DESCRIPTION:
Intake of carbohydrate-rich foods transiently increases blood glucose levels (known as postprandial glycaemia). Repeated high postprandial glucose responses are evidenced to dysregulate functional proteins, oxidative stress and pancreatic beta cell function; thus increasing the risk of diabetes and cardiovascular disease. Accordingly, meals that elicit a reduced, or more gradual, rise in blood glucose levels are desirable. Fruit polyphenols may help to limit the glucose excursion following a high carbohydrate meal. Previous research by our group has demonstrated that blackcurrant polyphenols significantly inhibited the average incremental area under the curve (T+0 to +30 min) of plasma glucose. Possible mechanisms include inhibition of intestinal enzymes and inhibition of intestinal glucose absorption by decreasing Sodium-glucose linked transporter 1 (SGLT-1) / Glucose transporter 2 (GLUT-2) glucose transporter activity. In vitro data suggests that citrus polyphenols may impact on carbohydrate metabolism by binding to starch molecules, however, effects on postprandial glycaemia are not yet known. Blackcurrants and citrus fruits have distinct polyphenol profiles and may therefore act on glucose homeostasis via different mechanisms. Blackcurrants are rich in anthocyanins and flavanols, whereas citrus fruits are rich in flavanones, hesperetin and naringenin. Theoretically, combining blackcurrant with citrus extracts may have synergistic effects.

The aim of this study is to investigate the effects of blackcurrant polyphenol extracts and citrus polyphenol extracts (and their combination), on postprandial glycaemia, insulinaemia and gastrointestinal hormone concentrations following a mixed carbohydrate test meal. It is hypothesised that blackcurrant and citrus extracts alone will inhibit glycaemia compared to placebo, a combination of the two will have a greater effect.

Study design: A randomised, controlled, double-blind, cross-over study will be conducted. Subjects will consume different drinks at 4 separate study visits. Drinks will contain either: blackcurrant extract (low dose), blackcurrant extract (high dose), citrus extract (low dose), blackcurrant and citrus extract (low dose + low dose), or placebo (no polyphenols). The study will utilise an incomplete block design. Subjects will consume the placebo drink and 3 out of 4 of the polyphenol-containing drinks during the study. At least a 7-day wash-out period will be required between study days. Baseline (fasted) blood samples will be taken in duplicate at T-10 min and T-5 min before consuming the test drink (T+0 min). Immediately following consumption of the drink, a mixed carbohydrate test meal will be consumed. Further blood samples will be collected at 10 min intervals for the first 30 min and then every 15 min until T+90 min and at T+120 min. Blood samples will be analysed for plasma glucose, insulin, glucose-dependent insulinotropic peptide (GIP), glucagon-like peptide 1 (GLP-1), peptide YY (PYY), C-peptide and nonesterified fatty acids (NEFA).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years
* Men and women
* Healthy (free of diagnosed diseases listed in the exclusion criteria)
* Body Mass Index 18-35 kg/m2
* Able to understand the information sheet and willing to comply with study protocol
* Able to give informed written consent

Exclusion Criteria:

* Those diagnosed with Phenylketonuria (PKU)
* Those with known or suspected food intolerances, allergies or hypersensitivity
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are breast feeding
* Participation in another clinical trial
* Those who have donated blood within 3 months of the screening visit and participants for whom participation in this study would result in having donated more than 1500 millilitres of blood in the previous 12 months.
* Full Blood Counts and Liver Function test results outside of the normal range.
* Current smokers, or reported giving up smoking within the last 6 months
* History of substance abuse or alcoholism
* Reported history of Cardiovascular disease, diabetes (or fasting glucose ≥ 7.1 mmol/L), cancer, kidney, liver or bowel disease, gastrointestinal disorder or use of drug likely to alter gastrointestinal function
* Unwilling to restrict consumption of specified high polyphenol foods for 48 h before the study
* Weight change >3kg in preceding 2 months
* Blood pressure ≥160/100 mmHg
* Total cholesterol ≥ 7.5 mmol/L; fasting triacylglycerol concentrations ≥ 5.0 mmol/L
* Medications that may interfere with the study: alpha-glucosidase inhibitors (acarbose: Glucobay), insulin sensitizing drugs (metformin: Glucophage, Glucophage SR, Eucreas, Janumet; thiazolidinediones: Actos, Competact), sulfonylureas (Daonil, Diamicron, Diamicron MR, Glibenese, Minodiab, Amaryl Tolbutamide), and lipid lowering drugs (statins, nicotinic acid, colestyramine anhydrous, ezetimibe, fibrates). Other medications should be reviewed by medical representative from KCL on a case by case basis.
* Nutritional supplements that may interfere with the study: higher dose vitamins/minerals (>200% Recommend Nutrient Intake), B vitamins, Vitamin C, calcium, copper, chromium, iodine, iron, magnesium, manganese, phosphorus, potassium and zinc. Subjects already taking vitamin or minerals at a dose around 100% or less up to 200% of the RNI, or evening primrose/algal/fish oil supplements will be asked to maintain habitual intake patterns, ensuring that they take them every day and not sporadically. They will be advised not to stop taking supplements or start taking new supplements during the course of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Postprandial glycaemia (iAUC 0-30 min) | 30 min
  The primary endpoint is iAUC 0-30 min for plasma glucose concentrations

SECONDARY OUTCOMES:
Postprandial glycaemia: iAUC 0-120 min | 120 min
  iAUC 0-120 min for plasma glucose concentrations
Postprandial glycaemia: iCmax | 120 min
  iCmax for plasma glucose concentrations
Postprandial glycaemia: Tmax | 120 min
  Tmax for plasma glucose concentrations
Postprandial glycaemia: absolute concentrations at specific time points | 120 min
  Absolute concentrations at specific time points, for plasma glucose concentrations
Postprandial insulinemia: iAUC 0-30 min | 30 min
  iAUC 0-30 min for serum insulin concentrations
Postprandial insulinemia: iAUC 0-120 min | 120 min
  iAUC 0-120 min for serum insulin concentrations
Postprandial insulinemia: iCmax | 120 min
  iCmax, for serum insulin concentrations
Postprandial insulinemia: Tmax | 120 min
  Tmax for serum insulin concentrations
Postprandial insulinemia: absolute concentrations at specific time points | 120 min
  Absolute concentrations at specific time points, for serum insulin concentrations
Postprandial C-peptide: iAUC 0-30 min | 30 min
  iAUC 0-30 min for plasma C-peptide concentrations
Postprandial C-peptide: iAUC 0-120 min | 30 min
  iAUC 0-120 min for plasma C-peptide concentrations
Postprandial C-peptide: iCmax | 120 min
  iCmax for plasma C-peptide concentrations
Postprandial C-peptide: Tmax | 120 min
  Tmax for plasma C-peptide concentrations
Postprandial C-peptide: Absolute concentrations at specific time points | 120 min
  Absolute concentrations at specific time points, for plasma C-peptide concentrations
Postprandial non-esterified fatty acids (NEFA): iAUC 0-30 min | 30 min
  iAUC 0-30 min for serum NEFA concentrations
Postprandial non-esterified fatty acids (NEFA): iAUC 0-120 min | 120 min
  iAUC 0-120 min for serum NEFA concentrations
Postprandial non-esterified fatty acids (NEFA): iCmax | 120 min
  iCmax for serum NEFA concentrations
Postprandial non-esterified fatty acids (NEFA): Tmax | 120 min
  Tmax for serum NEFA concentrations
Postprandial non-esterified fatty acids (NEFA): Absolute concentrations at specific time points | 120 min
  Absolute concentrations at specific time points, for serum NEFA concentrations
Postprandial blood glucose-dependent insulinotropic peptide (GIP): iAUC 0-30 min | 30 min
  iAUC 0-30 min for plasma GIP concentrations
Postprandial blood glucose-dependent insulinotropic peptide (GIP): iAUC 0-120 min | 120 min
  iAUC 0-120 min for plasma GIP concentrations
Postprandial blood glucose-dependent insulinotropic peptide (GIP): iCmax | 120 min
  iCmax, for plasma GIP concentrations
Postprandial blood glucose-dependent insulinotropic peptide (GIP): Tmax | 120 min
  Tmax for plasma GIP concentrations
Postprandial blood glucose-dependent insulinotropic peptide (GIP): Absolute concentrations at specific time points | 120 min
  Absolute concentrations at specific time points, for plasma GIP concentrations
Postprandial blood Glucagon-like peptide 1 (GLP-1): iAUC 0-30 min | 30 min
  iAUC 0-30 min for plasma GLP-1 concentrations
Postprandial blood Glucagon-like peptide 1 (GLP-1): iAUC 0-120 min | 120 min
  iAUC 0-120 min, for plasma GLP-1 concentrations
Postprandial blood Glucagon-like peptide 1 (GLP-1): iCmax | 120 min
  iCmax for plasma GLP-1 concentrations
Postprandial blood Glucagon-like peptide 1 (GLP-1): Tmax | 30 min
  Tmax for plasma GLP-1 concentrations
Postprandial blood Glucagon-like peptide 1 (GLP-1): Absolute concentrations at specific time points | 120 min
  Absolute concentrations at specific time points, for plasma GLP-1 concentrations
Postprandial blood peptide YY (PYY): iAUC 0-30 min | 30 min
  iAUC 0-30 min for plasma PYY concentrations
Postprandial blood peptide YY (PYY): iAUC 0-120 min | 120 min
  iAUC 0-120 minfor plasma PYY concentrations
Postprandial blood peptide YY (PYY): iCmax | 120 min
  iCmax for plasma PYY concentrations
Postprandial blood peptide YY (PYY): Tmax | 120 min
  Tmax for plasma PYY concentrations
Postprandial blood peptide YY (PYY): Absolute concentrations at specific time points | 120 min
  Absolute concentrations at specific time points, for plasma PYY concentrations

OTHER OUTCOMES:
Food diary (estimated/unweighed) | 7-days, collected at screening
  Habitual dietary intake analysis
VAS measures of the palatability of the study drink | 10 min following the test drink
  Descriptive statistics
VAS measures of mood, satiety and digestive comfort | 120 min
  Descriptive statistics
Buccal mouth swab | One off sample, collected at screening
  Future exploratory analysis of lactase activity via the derived allele at the European lactase persistence (LP) locus

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Hall, PhD, Principal Investigator — King's College London
Locations (1):
- Metabolic Research Unit, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castro-Acosta ML, Smith L, Miller RJ, McCarthy DI, Farrimond JA, Hall WL. Drinks containing anthocyanin-rich blackcurrant extract decrease postprandial blood glucose, insulin and incretin concentrations. J Nutr Biochem. 2016 Dec;38:154-161. doi: 10.1016/j.jnutbio.2016.09.002. Epub 2016 Sep 14. PMID 27764725
- [Derived] Pinto AM, Hobden MR, Brown KD, Farrimond J, Targett D, Corpe CP, Ellis PR, Todorova Y, Socha K, Bahsoon S, Haworth C, Marcel M, Nie X, Hall WL. Acute effects of drinks containing blackcurrant and citrus (poly)phenols and dietary fibre on postprandial glycaemia, gut hormones, cognitive function and appetite in healthy adults: two randomised controlled trials. Food Funct. 2023 Nov 13;14(22):10163-10176. doi: 10.1039/d3fo03085g. PMID 37902089